CLINICAL TRIAL: NCT00362869
Title: Pathogenicity of Enteroaggregative E. Coli in Adult Volunteers; Dose-Escalation Study
Brief Title: Enteroaggregative E.Coli (EAEC)
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: 02-209; UTHSC-H UCRC 1-5-03-023
Record Dates: First submitted 2006-08-10; First posted 2006-08-15 (Estimated); Last update posted 2016-12-26 (Estimated); Status verified 2010-04

CONDITIONS: Escherichia Coli Infections
Keywords: Enteroaggregative Escherichia coli, diarrhea, challenge
MeSH Terms: conditions — Escherichia coli Infections; Diarrhea | interventions — Levofloxacin; heat stable toxin (E coli)

ARMS (5):
- 1 (Experimental): Dosage 1X10^9 given orally in a sodium bicarbonate solution
  Interventions: Drug: Levofloxacin; Drug: Placebo; Biological: Enteroaggregative E. coli (EAEC)
- 2 (Experimental): Dosage 5X10^9 given orally in a sodium bicarbonate solution
  Interventions: Drug: Levofloxacin; Drug: Placebo; Biological: Enteroaggregative E. coli (EAEC)
- 5 (Placebo Comparator): Sodium bicarbonate placebo solution
  Interventions: Drug: Levofloxacin; Drug: Placebo
- 4 (Experimental): Dosage 5X10^10 given orally in a sodium bicarbonate solution
  Interventions: Drug: Levofloxacin; Drug: Placebo; Biological: Enteroaggregative E. coli (EAEC)
- 3 (Experimental): Dosage 1X10^10 given orally in a sodium bicarbonate solution
  Interventions: Drug: Levofloxacin; Drug: Placebo; Biological: Enteroaggregative E. coli (EAEC)

INTERVENTIONS:
Drug: Levofloxacin — Administered at a dose of 500 mg once a day for 3 days
Drug: Placebo — Sodium bicarbonate solution
Biological: Enteroaggregative E. coli (EAEC) — Dosages: 1X10^9, 5X10^9, 1X10^10, and 5X10^10 cfu; given in a sodium bicarbonate solution
  Arms: 1; 2; 3; 4

SUMMARY:
Enteroaggregative E. coli (EAEC) is a bacterium that can cause diarrhea. The purposes of this study are to: determine how much EAEC is needed to cause diarrhea in a healthy person, determine if a genetic factor is important in causing diarrhea, and to see how the body's defenses control EAEC. Participants include 25 healthy adults, ages 18-40. Volunteers will be assigned to 1 of 4 dose levels in groups of 5 volunteers each. One volunteer in each group will receive a sodium bicarbonate placebo solution. Volunteers will be admitted to the University Clinical Research Unit for up to 8 days. Volunteers will receive therapy with levofloxacin to treat the infection either once they develop diarrhea or at Day 5 if they remain asymptomatic. Study procedures will include saliva, blood, and fecal sample collection. An optional study procedure will include an intestinal biopsy. Participants will be involved in study related procedures for up to 223 days.

DETAILED DESCRIPTION:
Enteroaggregative Escherichia coli (EAEC) causes diarrhea in travelers from industrialized nations to developing countries, children of developing countries, and patients with HIV. Although infection responds to antibiotic therapy, increasing antibiotic resistance and the widespread nature of the infection limit the utility of antibiotics. The development of an EAEC-specific vaccine would be useful in the prevention of travel-associated EAEC diarrhea and in the decrease of EAEC-associated mortality in young children in the US and of developing countries. The first objective of the study is to perform a dose-escalation study of EAEC 042 infectivity in healthy adult volunteers who are high producers of IL-8 and seronegative to EAEC. The study will identify the dose of EAEC 042 needed for future studies on EAEC 042 such as phase I-II EAEC vaccine studies. The second objective of the study is to identify the humoral, secretory, and cellular immune response to EAEC 042 specific antigens that are associated with EAEC infection. Study participants will include 25 healthy volunteers, ages 18-40, from the greater Houston area. Study participants will be assigned to 1 of 4 possible dose levels in groups of 5 volunteers each. Each study group will consist of 4 volunteers receiving EAEC and 1 volunteer receiving a sodium bicarbonate placebo solution. Safety data and results will be reviewed by the safety monitoring committee before beginning the next highest dose group. If a dose results in at least 3 of the 4 infected volunteers of a given group, the next highest dose will not be administered. Instead, the concentration will be repeated for validation of the dose. Healthy volunteers will be screened as outpatients for the presence of the -251 AA SNP genotype in the IL-8 gene promoter. Once a volunteer has been screened and determined to be eligible to participate in the study, the volunteer will sign a consent form and be admitted at the University Clinical Research Unit. The volunteer will ingest a determined concentration of EAEC 042 or placebo and be observed for symptoms of infection. All volunteers will receive therapy with levofloxacin to eradicate the infection either once they develop diarrhea or at Day 5 if they remain asymptomatic. Volunteers will be discharged from the hospital on Day 7+/-1. Saliva, blood, and feces will be collected for secretory, humoral, and cellular immune responses to EAEC. An optional procedure will consist of obtaining jejunal and colonic biopsies prior to challenge (Day -13±2) and Days 4±1 and 24±3 post challenge. Volunteer participation in endoscopy studies will be optional and will not be a requirement for the rest of the study. The primary endpoints of the study include: diarrheal illness after exposure to EAEC, shedding of EAEC after exposure, and IgG and secretory IgA (slgA) seroconversion to EAEC dispersin. The secondary endpoints of the study include: increase in fecal markers of intestinal inflammation including cytokines and lactoferrin and description of the jejunal and colonic immune response to EAEC infection.

ELIGIBILITY:
Inclusion Criteria:

* Sign an Institutional Review Board-approved consent prior to any study-related activities.
* Initiate screening 21± 7 days prior to admission or enrollment.
* Must accomplish all laboratory and diagnostic examinations at 21± 7 days prior to admission or enrollment.
* Be at least 18 years of age but not older than 40 years of age at the time of enrollment.
* Be otherwise healthy with a stable address and telephone where the volunteer can be contacted.
* Be able to read and write English.
* Possess a social security number in order to receive compensation.
* Female participants must have a negative serum pregnancy test at screening and a negative urine pregnancy test on the morning of the challenge and use effective birth control during the entire study period. Methods of effective birth control include: complete abstinence, the use of a licensed hormonal method, intrauterine device, barrier method plus spermicide, or having sexual relations exclusively with a vasectomized partner. Appropriate barrier methods include condoms, cervical sponge, and diaphragm. Females who are not of childbearing potential are defined as those who are physiologically incapable of becoming pregnant, including any female with tubal ligation or who is postmenopausal. For purposes of this study, postmenopausal status will be defined as absence of menses for at least 1 year.
* Be seronegative for antibodies to dispersin.
* Have normal laboratory screening values including a white blood cell (WBC) count, hemoglobin, hematocrit, platelets, blood urea nitrogen, glucose, creatinine, alanine aminotransferase (ALT), aspartate aminotransferase (AST), quantitative immunoglobulins, T cell subsets (CD4 and CD8), urinalysis.
* Have normal chest x-ray and electrocardiogram.
* Have negative serologies for HIV, hepatitis B virus (HBV), and hepatitis C virus (HCV), and a negative rapid plasma reagin (RPR).
* Have a negative stool examination for pathogenic ova and pathogenic parasites, and bacterial enteropathogens (EAEC, Salmonella, Shigella, Campylobacter).
* Have the -251 AA IL-8 genotype.

Exclusion Criteria:

* Has acute or chronic medical illness (i.e., renal or hepatic disease, hypertension, diabetes mellitus, coronary artery disease, malnutrition, obesity (body mass index >30 kg/m2), HIV, corticosteroid use, cancer or receiving chemotherapy, chronic debilitating illness, syphilis).
* Has used antibiotics within 7 days of challenge.
* Has used medications or drugs, including over-the-counter medications such as decongestants, antacids (calcium carbonate or aluminum-based antacids, H2 blockers), anti-diarrheal medications (such as bismuth subsalicylate or loperamide), antihistamines within 7 days of challenge.
* Has a history of chronic gastrointestinal illness, intra-abdominal surgery, chronic functional dyspepsia, chronic gastroesophageal reflux, documented peptic ulcer disease, gastrointestinal hemorrhage, gallbladder disease, inflammatory bowel disease (Crohn's and ulcerative colitis), diverticulitis, irritable bowel syndrome or frequent diarrhea.
* Has a history any of the following psychiatric illness(es):
* Depression not controlled with current drug therapy or involving institutionalization
* Schizophrenia or psychosis
* Suicide attempt.
* Has a history of or current alcohol or illicit drug abuse.
* Is unable to remain as an inpatient in the University Clinical Research Unit for up to 8 days.
* Has a known hypersensitivity to latex, heparin, opiates, antiemetics, benzodiazepines, lidocaine, magnesium citrate, or Fleet enema.
* Has a known hypersensitivity to antibiotics that could be used to treat EAEC infection including fluoroquinolones, amoxicillin, cephalosporins or rifaximin.
* Has serum antibodies to EAEC dispersin.
* Recently traveled to a developing country (within 6 months).
* Has household contacts who are less than 4 years of age or more than 80 years of age.
* Has household contacts that are infirmed or immunocompromised due to any of the following reasons:
* Corticosteroid therapy
* HIV infection
* Cancer chemotherapy
* Other chronic debilitating diseases.
* Works as health care personnel with direct patient care.
* Works in a day care center for children or the elderly.
* Is a food handler.
* Has factors that, in the opinion of the investigator or research personnel, would interfere with the study objectives or increase the risk to the volunteer or his contacts.
* Is currently participating in a clinical study or had receipt of an investigational drug in the past 30 days.
* Is pregnant or has a risk of pregnancy or is lactating.
* Has current excessive use of alcohol or drug dependence.
* Has evidence of impaired immune function.
* Has a new positive reaction to purified protein derivative (PPD) (volunteers who are known to be PPD positive that have a negative chest x-ray and have received isoniazid prophylaxis will be eligible).
* Has a stool culture that demonstrates the presence of pathogenic ova, pathogenic parasites, or bacterial enteropathogens (EAEC, Salmonella, Shigella, and Campylobacter), or that is devoid of normal flora.
* Has self-reported lactose or soy intolerance or allergy
* Is a smoker and cannot stop smoking for the duration of the inpatient study.
* Has abnormal lab results for screening beyond the normal range as defined below:

Hematology Hemoglobin: 13-15.0 gm/dL (Females) 14.5-17.0 gm/dL (Males) Hematocrit: 37-46 % (Females) 40-52 % (Males) Platelet count: 140,000-415,000 per mm3 WBC count: 4,000-10,500 per mm3 Neutrophils: 40-74 % or 1,800-7,800 per mm3 Lymphocytes: 14-26 % or 700-4,500 per mm3 Monocytes: 4-13 % or 100-1,000 per mm3 Eosinophils: 0-7 % or 0-400 per mm3 Basophils: 0-3 % or 0-200 per mm3

Chemistry BUN 5-25 mg/dL Creatinine 0.5-1.4 mg/dL Glucose (fasting) 69-99 mg/dL ALT 0-40 U/L AST 0-40 U/L

Immunology IgG: 596-1584 mg/dL IgA: 71-350 mg/dL IgM: 35-213 mg/dL CD4 T cells: 660-1500 cells/mcl CD8 T cells: 360-850 cells/mcl

Urinalysis Urine color: Yellow Turbidity: Clear pH: 5.0-8.0 Protein: Negative Sp. Gravity: 1.003-1.030 Glucose: Negative WBC: 0-2 Cells per HPF RBC: 0 Cells per HPF Bacteria: Rare Ketones: Negative The urinalysis will initially be evaluated for the quality of collection. If urinalysis is found to be poorly collected and demonstrates the presence of squamous epithelial cells and bacteria, results will not be used and a repeat urinalysis will be requested. In the case of menstruating women, the urinalysis collection will be postponed temporarily. A urinalysis may also be repeated once if traces of bile, protein, trace ketones, or Hb are identified. In the case of a properly collected urinalysis, the presence of leukocyte esterase glucose, or nitrates will exclude the participation of the subject.

* Occult blood (Hemoccult) positive stools on admission to the CRU.
* Develops gastrointestinal symptoms including nausea, vomiting, anorexia, abdominal pain, cramping, bloating, excessive gas or flatulence, diarrhea, constipation, urgency or tenesmus between the screening period and prior to challenge.
* Develops a febrile illness during the period of time screening period and prior to challenge.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 5 (Actual)
Dates: Start 2008-02; Primary Completion 2008-08 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Development of diarrhea defined as passage of one diarrheal stool containing at least 300 mL or 2 or more stools totaling 200 mL or greater passed during a 48-hour period within 96 hours after challenge. | Assessed daily during the inpatient portion of the study

SECONDARY OUTCOMES:
Increases in individual markers of inflammation: fecal leukocytes, lactoferrin and pro-inflammatory cytokines. | At the conclusion of the challenge studies, once all specimens have been collected.
Proportion of subjects who receive rescue antibiotic therapy (defined as the initiation of antibiotic therapy when the primary outcome criteria listed above is met). | Assessed daily during the inpatient portion of the study, Days 0-8
Secretory IgA and humoral IgG response to homologous administered strain; expressed in titers. | At the conclusion of the challenge studies, once all specimens have been collected.
Total volume of unformed stools passed during 5 days of study. | Assessed daily during the inpatient portion of the study
Positive excretion of the administered test strain and number of days of excretion before antimicrobial is administered. | Assessed daily during the inpatient portion of the study
Development of mild diarrhea defined as passage of any number of stools categorized as loose or watery but of less than 200 mL in addition to a complaint of one or more enteric symptoms. | Assessed daily during the inpatient portion of the study

CONTACTS AND LOCATIONS:
Locations (1):
- University of Texas Health Science Center, Houston, Texas, United States